CLINICAL TRIAL: NCT06468657
Title: Evaluation of the Impact of Ejection Fraction on Clinical Outcomes in Patients Undergoing Cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ejection fraction
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low | interventions — Mortality; Vasoconstrictor Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- reduced ejection fraction: EF below 50
  Interventions: Other: mortality rates
- preserved ejection fraction: EF above 50
  Interventions: Other: mortality rates

INTERVENTIONS:
Other: mortality rates — mortality rates
  Other Names: vasopressor/inotropic agent needs; transfusion needs; perioperative arrhythmias; intensive care stay

SUMMARY:
This study evaluates the impact of ejection fraction (EF) on clinical outcomes in patients undergoing cardiovascular surgeries, specifically coronary artery bypass grafting (CABG) and heart valve replacement. It spans surgeries performed between 2012 and 2022 at Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital. Patients are categorized into two groups based on their preoperative EF: those with preserved EF (≥50%) and those with reduced EF (<50%).

The primary aim is to assess how EF affects postoperative morbidity, mortality, hospital stay, and complications. Secondary aims include evaluating the development of postoperative arrhythmias, the need for vasopressors and inotropes, and transfusion requirements.

Data will be collected retrospectively from hospital records and electronic health systems. The study's findings are expected to provide insights into tailored perioperative and postoperative management strategies for patients with varying EF levels, ultimately improving clinical outcomes.

DETAILED DESCRIPTION:
Primary Objective The primary objective of this study is to evaluate the impact of ejection fraction (EF) on clinical outcomes in patients undergoing cardiovascular surgery. Specifically, the study aims to analyze the effects of EF on postoperative morbidity and mortality rates, length of hospital stay, and postoperative complications.

Secondary Objectives Secondary objectives include assessing the development of arrhythmias in the postoperative period, the need for vasopressors and inotropes, and the requirement for transfusions.

Scope of the Study Time Frame The study will encompass cardiovascular surgeries performed between 2012 and 2022. This time frame is selected to obtain a sufficient data set and evaluate long-term outcomes.

Research Center The study will be conducted at Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital. Patient data from cardiovascular surgeries performed at this center will be analyzed.

Patient Population The study will include all patients who underwent cardiovascular surgery within the specified time frame and had preoperative ejection fraction (EF) measurements.

Study Design Group Formation

Patients will be divided into two main groups based on their preoperative EF values:

Preserved EF Group: Patients with an EF of 50 or above. Reduced EF Group: Patients with an EF below 50. Data to be Examined

The following postoperative data will be examined and compared between the two groups:

Development of Postoperative Arrhythmias: Whether patients develop arrhythmias in the postoperative period.

Vasopressor Requirement: The need for vasopressors in the postoperative period. Inotrope Requirement: Whether patients require inotropic support postoperatively.

Transfusion Requirement: The need for blood transfusions in the postoperative period.

Mortality: Survival rates of patients following surgery. Need for Revision Surgery: Whether patients require additional surgical interventions postoperatively.

Length of Stay in ICU: Duration of patients' stay in the intensive care unit. Total Hospital Stay: Overall length of hospital stay. Data Collection Method Data will be retrospectively collected from hospital records and electronic health record (EHR) systems.

This structured approach aims to comprehensively evaluate the clinical outcomes of patients with varying levels of ejection fraction undergoing major cardiovascular surgeries, thereby providing insights that can enhance patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients aged 18 years and older.
* Cardiovascular Surgery: Patients who have undergone cardiovascular surgeries such as coronary artery bypass grafting (CABG), valve surgery, aortic surgery, etc.
* Ejection Fraction (EF): Patients with documented EF measurements.

Exclusion Criteria:

* Age: Patients under 18 years of age.
* Non-Surgical Interventions: Patients undergoing procedures other than cardiovascular surgery.
* Incomplete Data: Patients without documented EF measurements or with missing clinical data.
* Pregnancy: Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 210 patients who underwent cardiovascular surgery at Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital and had their ejection fraction (EF) measured in the preoperative period will be included in the study.
Sampling Method: Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days
  mortality in 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No